CLINICAL TRIAL: NCT03983408
Title: Impact of Korean Red Ginseng on Fatigue in Patients With Rheumatic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Collaborators: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Yoon-Kyoung Sung, Professor, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUHRD-SPE-19-01
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Sjögren's Syndrome; Rheumatic Diseases; Korean Red Ginseng
Keywords: Sjögren's Syndrome; Korean Red Ginseng
MeSH Terms: conditions — Sjogren's Syndrome; Rheumatic Diseases | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation concealment for first 12 weeks is maintained; all participants are provided with KRG during during another 12 weeks for the open-label extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KRG group (Active Comparator): * Enrollment: 60 patients
  * Drug: Korean Red Ginseng (KRG) 2,000 mg/day for total 24 weeks (2 Korean Red Ginseng extract tablet twice a day, ginsenoside Rg1+Rb1+Rg3 7.0 mg/g per each tablet)
  Interventions: Dietary Supplement: Korean Red Ginseng
- Placebo group (Placebo Comparator): * Enrollment: 60 patients
  * Drug: Placebo for 12 weeks, following Korean Red Ginseng 2,000mg/day for another 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — Participants are provided with 2 Korean Red Ginseng extract tablets twice a day for total 24 weeks.
  Other Names: KRG
  Arms: KRG group
Dietary Supplement: Placebo — Placebo tablets, made of corn starch and cellulose, are manufactured to mimic KRG tablets. Participants are parovided with 2 placebo tablets twice a day for first 12 weeks, following Korean Red Ginseng extract tablets twice a day for another 12 weeks.
  Arms: Placebo group

SUMMARY:
The objective of a randomized, double-blind, placebo-controlled trial and open-label extension study is to figure out the impact of Korean Red Ginseng (KRG) on fatigue in patients with rheumatic diseases.

DETAILED DESCRIPTION:
Primary objective

: Improvement of fatigue after using KRG in patients with rheumatic diseases according to

Secondary objectives

1. Improvement of dryness after using KRG in patients with rheumatic diseases according to EULAR Sjögren's syndrome disease activity index (ESSDAI)
2. Improvement of quality of life after using KRG in patients with rheumatic diseases according to EuroQol 5 dimensions questionnaire (EQ-5D)

The study population will be adult patients with rheumatic diseases, especially primary or secondary Sjögren's syndrome who have experienced dryness for more than 3 months. Participants are ramdomly assigned to KRG and placebo group and they are using KRG or placebo for the first 12 weeks. After 12 weeks, the concealment of allocation is lifted and all patients are provided with KRG for next 12 weeks with open-label extension study

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet for Classification Criteria for Sjögren's syndrome
* Patients who have experienced fatigue for over 3 months
* Patients aged ≥ 19 and <75
* Patients who provide a written consent of participating in this study.

Exclusion Criteria:

* Patients who have experienced hypersensitivity or adverse events to Korean Red ginseng
* Patients who used dietary supplements containing KRG during recent 2 months
* Patients who are pregnant or breast-feeding
* Patients who use oral glucocorticoids or opioids continuously
* Patients who had other comorbidities which could lead to fatigue as symptoms including chronic kidney disease, chronic liver disease, endocrine disoders, malignancy, or depression.
* Patients having fibromyalgia or chronic fatigue syndrome
* Patients who presented abnormal laboratory findings at the time of enrollment White blood cell (WBC) ≤ 3.5 x 10^9/L or, Hemoglobin (Hb) ≤ 8.5 g/dL or, Platelet (PLT) ≤ 100 x 10^9/L or, Serum creatinine (Cr) ≥ 2.0 mg/dL or, Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥ 2.5 times of upper limits of normal

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The Functional Assessment of Chronic Illness-Fatigue (FACIT-F, total score ranged 0 to 52, higher scores respresent less fatigue) | 12 weeks
  Improvement of FACIT-F after using KRG

SECONDARY OUTCOMES:
Visual analogue scale-Fatigue (VAS-F, total score ranged 0 [fatigued not at all] to 100 [extremely fatigued]) | 12 weeks
  Improvement of FACIT-VAS after using KRG
ESSDAI (The EULAR Sjögren's syndrome [SS] disease activity index, total score ranged 0 to 123, higher scroes indicate severe systemic disease activity) | 12 weeks
  Improvement of ESSDAI after using KRG
EuroQol 5 dimensions questionnaire (EQ-5D, a person's health status is defined by a 5-digit number, ranging from 11111 [having no problems in all dimensions] to 33333 [having extreme problems in all dimensions]) | 12 weeks
  Improvement of EQ-5D after using KRG

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Kyoung Sung, MD, PhD, MPH, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD is not shared with other researchers

REFERENCES:
- [Background] Cho SK, Kim D, Yoo D, Jang EJ, Jun JB, Sung YK. Korean Red Ginseng exhibits no significant adverse effect on disease activity in patients with rheumatoid arthritis: a randomized, double-blind, crossover study. J Ginseng Res. 2018 Apr;42(2):144-148. doi: 10.1016/j.jgr.2017.01.006. Epub 2017 Jan 20. PMID 29719460